CLINICAL TRIAL: NCT02681328
Title: Randomized Trial Comparing Performance of Molecular Markers for Indeterminate Thyroid Nodules
Status: Active, not recruiting | Type: Observational
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 16-000055
Record Dates: First submitted 2016-02-10; First posted 2016-02-12 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Thyroid
MeSH Terms: conditions — Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Afirma GEC: single molecular test GEC of collected tissue
  Interventions: Other: Afirma GEC
- ThyroSeq v.2: single molecular test ThyroSeq v.2 of collected tissue
  Interventions: Other: ThyroSeq v.2
- Afirma GSC: single molecular test GSC of collected tissue
  Interventions: Other: Afirma GSC
- ThyroSeq v.3: single molecular test ThyroSeq v.3 of collected tissue
  Interventions: Other: ThyroSeq v.3

INTERVENTIONS:
Other: Afirma GEC — Afirma GEC molecular test on collected thyroid tissue
  Groups: Afirma GEC
Other: ThyroSeq v.2 — ThyroSeq v.2 molecular test on collected thyroid tissue
  Groups: ThyroSeq v.2
Other: Afirma GSC — Afirma GSC molecular test on collected thyroid tissue
  Groups: Afirma GSC
Other: ThyroSeq v.3 — ThyroSeq v.3 molecular test on collected thyroid tissue
  Groups: ThyroSeq v.3

SUMMARY:
The purpose of this study is to compare the performance of Afirma GSC and ThyroSeq v.3 in indeterminate thyroid nodules to determine which test can allow more patients to avoid unnecessary surgery and preserve quality of life. In the initial phase of this study, the performance of Afirma GEC and ThyroSeq v.2 were compared.

DETAILED DESCRIPTION:
1. All patients undergoing thyroid FNA within the UCLA Health System will be randomized at the time of FNA to a single molecular test (GSC or ThyroSeq v.3). In the previous phase of the study, patients were randomized to the previous versions of a single molecular test (GEC or ThyroSeq v.2).
2. During the FNA, a sample will be collected for the molecular test.
3. If the cytology results are indeterminate (Bethesda categories 3 or 4), the molecular test will be reflexively sent off.
4. We will help patients with indeterminate thyroid nodules to establish care with an endocrinologist, if they do not already have one. The physicians will make treatment recommendations using best practices and incorporating the results of the molecular test. We anticipate that most patients with a positive molecular test will undergo surgery, while the majority with a negative test will be surveiled.
5. Patients who undergo surgery will have histopathologic evaluation of the thyroid, which will determine whether the index thyroid nodule was benign or malignant.
6. Patients who do not undergo surgery will have a followup ultrasound at 6 and 12 months, or sooner at the discretion of the treating physician.
7. We will assess thyroid-specific quality of life at baseline (following initial diagnosis of an indeterminate thyroid nodule) and during followup (at 6 and 12 months) using the short version of Thyroid-Related Patient-Reported Outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a thyroid nodule who have a thyroid biopsy performed at UCLA health will be eligible for the study and consented if they agree to participate.
* Patients who have an indeterminate FNA biopsy result (Bethesda category 3 or 4) will be enrolled in the study if they agree to participate.

Exclusion Criteria:

* Patients who do not have an indeterminate biopsy result (either patients who have a benign, insufficient, or malignant result).

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing thyroid fine needle aspiration (FNA) within the University of California, Los Angeles (UCLA) Health System
Sampling Method: Non-Probability Sample
Enrollment: 328 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Afirma GEC vs. ThyroSeq v.2 in indeterminate thyroid nodules post best practices surgery | 12 months. [This phase of the study is now completed]
  compare the performance of Afirma GEC and ThyroSeq v.2 in indeterminate thyroid nodules to determine which test can allow more patients to avoid unnecessary surgery and preserve quality of life. (5) Patients who undergo surgery will have histopathologic evaluation of the thyroid, which will determine whether the index thyroid nodule was benign or malignant.
2. Afirma GSC vs. ThyroSeq v.3 in indeterminate thyroid nodules post best practices surgery | 12 months.
  compare the performance of Afirma GSC and ThyroSeq v.3 in indeterminate thyroid nodules to determine which test can allow more patients to avoid unnecessary surgery and preserve quality of life. (5) Patients who undergo surgery will have histopathologic evaluation of the thyroid, which will determine whether the index thyroid nodule was benign or malignant.

SECONDARY OUTCOMES:
Avoidance of unnecessary surgeries | 12 months
  Determine the number of unnecessary surgeries avoided based on the number of false-positive test results, and assess whether this translated into improved quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Masha Livhits, MC, Principal Investigator — Visiting Assistant Professor
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cibas ES, Ali SZ; NCI Thyroid FNA State of the Science Conference. The Bethesda System For Reporting Thyroid Cytopathology. Am J Clin Pathol. 2009 Nov;132(5):658-65. doi: 10.1309/AJCPPHLWMI3JV4LA. PMID 19846805
- [Background] Lee L, How J, Tabah RJ, Mitmaker EJ. Cost-effectiveness of molecular testing for thyroid nodules with atypia of undetermined significance cytology. J Clin Endocrinol Metab. 2014 Aug;99(8):2674-82. doi: 10.1210/jc.2014-1219. Epub 2014 Mar 31. PMID 24684467
- [Background] Alexander EK, Kennedy GC, Baloch ZW, Cibas ES, Chudova D, Diggans J, Friedman L, Kloos RT, LiVolsi VA, Mandel SJ, Raab SS, Rosai J, Steward DL, Walsh PS, Wilde JI, Zeiger MA, Lanman RB, Haugen BR. Preoperative diagnosis of benign thyroid nodules with indeterminate cytology. N Engl J Med. 2012 Aug 23;367(8):705-15. doi: 10.1056/NEJMoa1203208. Epub 2012 Jun 25. PMID 22731672
- [Background] Nikiforov YE, Carty SE, Chiosea SI, Coyne C, Duvvuri U, Ferris RL, Gooding WE, LeBeau SO, Ohori NP, Seethala RR, Tublin ME, Yip L, Nikiforova MN. Impact of the Multi-Gene ThyroSeq Next-Generation Sequencing Assay on Cancer Diagnosis in Thyroid Nodules with Atypia of Undetermined Significance/Follicular Lesion of Undetermined Significance Cytology. Thyroid. 2015 Nov;25(11):1217-23. doi: 10.1089/thy.2015.0305. Epub 2015 Sep 10. PMID 26356635
- [Background] Wu JX, Lam R, Levin M, Rao J, Sullivan PS, Yeh MW. Effect of malignancy rates on cost-effectiveness of routine gene expression classifier testing for indeterminate thyroid nodules. Surgery. 2016 Jan;159(1):118-26. doi: 10.1016/j.surg.2015.05.035. Epub 2015 Oct 2. PMID 26435428
- [Background] Wu JX, Young S, Hung ML, Li N, Yang SE, Cheung DS, Yeh MW, Livhits MJ. Clinical Factors Influencing the Performance of Gene Expression Classifier Testing in Indeterminate Thyroid Nodules. Thyroid. 2016 Jul;26(7):916-22. doi: 10.1089/thy.2015.0505. Epub 2016 Jun 9. PMID 27161519
- [Derived] Hu TX, Nguyen DT, Patel M, Beckett K, Douek M, Masamed R, Rhyu J, Kim J, Tseng CH, Yeh MW, Livhits MJ. The Effect Modification of Ultrasound Risk Classification on Molecular Testing in Predicting the Risk of Malignancy in Cytologically Indeterminate Thyroid Nodules. Thyroid. 2022 Aug;32(8):905-916. doi: 10.1089/thy.2021.0659. Epub 2022 Jun 23. PMID 35611970
- [Derived] Zhu CY, Donangelo I, Gupta D, Nguyen DT, Ochoa JE, Yeh MW, Livhits MJ. Outcomes of Indeterminate Thyroid Nodules Managed Nonoperatively after Molecular Testing. J Clin Endocrinol Metab. 2021 Mar 8;106(3):e1240-e1247. doi: 10.1210/clinem/dgaa887. PMID 33394039
- [Derived] Livhits MJ, Zhu CY, Kuo EJ, Nguyen DT, Kim J, Tseng CH, Leung AM, Rao J, Levin M, Douek ML, Beckett KR, Cheung DS, Gofnung YA, Smooke-Praw S, Yeh MW. Effectiveness of Molecular Testing Techniques for Diagnosis of Indeterminate Thyroid Nodules: A Randomized Clinical Trial. JAMA Oncol. 2021 Jan 1;7(1):70-77. doi: 10.1001/jamaoncol.2020.5935. PMID 33300952
- [Derived] Livhits MJ, Kuo EJ, Leung AM, Rao J, Levin M, Douek ML, Beckett KR, Zanocco KA, Cheung DS, Gofnung YA, Smooke-Praw S, Yeh MW. Gene Expression Classifier vs Targeted Next-Generation Sequencing in the Management of Indeterminate Thyroid Nodules. J Clin Endocrinol Metab. 2018 Jun 1;103(6):2261-2268. doi: 10.1210/jc.2017-02754. PMID 29590358